CLINICAL TRIAL: NCT05143138
Title: Real-World Data Collection of the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis When Used as a Bridging Stent With Branched and Fenestrated Endografts in the Treatment of Aortic Aneurysms Involving the Renal-Mesenteric Arteries
Acronym: EMBRACE
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VBX 21-04
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysm; Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- fEVAR: Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent in conjunction with a fenestrated stent graft to allow endovascular aneurysm repair
  Interventions: Device: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis
- bEVAR: Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent in conjunction with a branched stent graft to allow endovascular aneurysm repair
  Interventions: Device: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis
- fEVAR and bEVAR: Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent in conjunction with a branched and fenestrated stent graft to allow endovascular aneurysm repair
  Interventions: Device: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis

INTERVENTIONS:
Device: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis — Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent

SUMMARY:
Multicenter, single-arm retrospective and prospective registry is being conducted to confirm the clinical performance and safety of GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis when used as a Bridging Stent with Branched and Fenestrated Endografts in the Treatment of Aortic Aneurysms Involving the Renal-Mesenteric Arteries.

DETAILED DESCRIPTION:
Up to 15 sites in Europe will be required to enroll a minimum of 220 patients that have had treatment with GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis when used as a Bridging Stent with Branched and Fenestrated Endografts in the Treatment of Aortic Aneurysms Involving the Renal-Mesenteric Arteries.

The registry procedures consist of two phases, retrospective phase and prospective phase.

The retrospective phase consists only of the collection of retrospective data (baseline, treatment and FU data) from the source documents available at the site from the time of the treatment until the enrollment date (ICF signature).

The prospective phase consists in collection of follow-up visits from the enrollment up to 5 years. The FU data collected prospectively can change from subject to subject depending on the index procedure date. Diagnostic imaging, treatment interventions, and follow up will be determined by physicians based on clinical practice standards.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent in conjunction with a branched/fenestrated stent graft to allow endovascular aneurysm repair from 31 December 2021 until 01 January 2017
2. Age ≥18 years at the time of implant
3. Provision of informed consent by the patient or next of kin/legal representative (for deceased patients at registry entry, unless a waiver was granted), according to local regulations.

Exclusion Criteria:

1. Patient treated for ruptured aneurysm or who were otherwise hemodynamically unstable at the time of the procedure
2. Patient treated for acute or sub-acute dissection, <90 days from onset of symptoms
3. Patient treated using physician-modified endovascular grafts
4. Patient intended to be treated with chimney, periscope, octopus, sandwich technique per the pre-treatment case plan
5. At the time of treatment, patient had known coagulation disorders including hypercoagulability that were not amenable to treatment
6. Patient was pregnant at the time of treatment.
7. Participation in another drug or device investigational study within one year of device implant, that can confound the registry endpoints.
8. Patient had known or suspected systemic infection (including treatment for mycotic aneurysm) at the time of implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry has been designed with broad eligibility criteria to capture real-world data about GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis used as a Bridging Stent in conjunction with a branched/fenestrated stent graft to allow endovascular aneurysm repair.
  Patients will be identified from hospital database.
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Bertoglio, Prof, Principal Investigator — spedali civili brescia
Locations (14):
- Denmark (2):
  - Aarhus University, Aarhus
  - Rigshospitalet, Copenhagen
- Italy (4):
  - IRCCS Ospedale Policlinico San Martino, Genova
  - "Vita-Salute" San Raffaele University I.R.C.C.S Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Complesso Ospedaliero San Giovanni Addolorata, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Roma
- AMC, Meibergdreef 9, Amsterdam, Netherlands
- Norway (3):
  - Haukeland Universitetssjukehus, Bergen
  - UNN Tromsø, Tromsø
  - St. Olavs Hospital, Trondheim
- Spain (2):
  - Hospital Clínico Universitario San Cecilio, Granada
  - Hospital Clinico San Carlos, Madrid
- Sweden (2):
  - Skane University Hospital, Malmo
  - Uppsala University Hospital, Uppsala

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 259 patients enrolled and divided as follows: 136 subjects in the BEVAR cohort, 92 in the FEVAR cohort and 31 in the MIXED cohort Fourteen investigators at 14 sites participated in the registry within 6 European countries. All the 14 sites are still active and enrolled subjects.
Period: Overall Study
Arm/Group | fEVAR | bEVAR | fEVAR and bEVAR
Started | 92 | 136 | 31
Completed (End of 1 year analysis window (POD 455).) | 84 | 96 | 30
Not Completed | 8 | 40 | 1
Not completed — Death | 5 | 35 | 1
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — withdrawal | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | fEVAR | bEVAR | fEVAR and bEVAR | Total
Number analyzed (Participants) | 92 | 136 | 31 | 259
Age, Continuous [Median (Full Range); unit: Years] | 74 [45 to 87] | 74 [28 to 89] | 72 [32 to 86] | 74 [28 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 37 | 14 | 63
  Male | 80 | 99 | 17 | 196
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 11 | 21 | 0 | 32
  Sweden | 13 | 18 | 7 | 38
  Norway | 22 | 1 | 7 | 30
  Denmark | 19 | 19 | 6 | 44
  Italy | 16 | 62 | 5 | 83
  Spain | 11 | 15 | 6 | 32
Serum Creatinine [Median (Full Range); unit: mg/dL] — Serum Creatinine, mg/dL
  mg/dL | 1.1 [0.4 to 6.4] | 1.1 [0.5 to 6.4] | 0.9 [0.5 to 2.0] | 1.1 [.4 to 6.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Vessel Patency
Description: Uninterrupted patency with no occlusion or procedure performed to maintain patency on the VBX Stent Graft or native target vessel. Interventions intended to treat endoleak or stent disconnection do not count as loss of primary patency. Binomial proportions were calculated at 12 month follow-up.
Time Frame: 12 months
Population: Study endpoints were planned and calculated for the two primary cohorts only. Subjects that are not discontinued prior to 1 year window and with imaging within 1 year window.
Measure: Count of Participants; unit: Participants
Arm/Group | fEVAR | bEVAR
Number analyzed (Participants) | 79 | 90
Participants | 78 | 84

ADVERSE EVENTS:
Time Frame: 1 year adverse events for primary cohorts. Time period is up to and including day 365, which is different than study analysis windows.
Description: Serious Adverse Event: Any adverse event that led to any of the following:
  1. death
  2. serious deterioration in the health of the subject, users, or other persons as defined by one or more of the following:
  3. fetal distress, fetal death, or a congenital abnormality, or birth defect including physical or mental impairment
Groups:
- fbEVAR: Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent in conjunction with a fenetrated or branched stent graft to allow endovascular aneurysm repair
  GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis: Patients treated with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis as a Bridging Stent
Arm/Group | fEVAR | bEVAR | fbEVAR
All-Cause Mortality (participants affected / at risk) | 5/92 | 35/136 | 1/31
Serious Adverse Events (participants affected / at risk) | 44/92 | 89/136 | 21/31
Other Adverse Events (participants affected / at risk) | 6/92 | 7/136 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | fEVAR (N=92) | bEVAR (N=136) | fbEVAR (N=31)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Decompensated heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ischemic heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
NSTEMI (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right heart failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
STEMI (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Bleeding duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bleeding gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bowel ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bowel ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paralytic ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Superior mesenteric artery dissection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fever of unknown origin (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hyposthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
In-stent arterial stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiorgan failure (General disorders) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Stent thrombosis (General disorders) | 0 (0) | 1 (2) | 0 (0)
Stent-graft endoleak type IA (General disorders) | 0 (0) | 2 (2) | 1 (1)
Stent-graft endoleak type IB (General disorders) | 4 (4) | 2 (2) | 0 (0)
Stent-graft endoleak type IC (General disorders) | 2 (2) | 8 (8) | 2 (3)
Stent-graft endoleak type II (General disorders) | 1 (1) | 7 (10) | 3 (3)
Stent-graft endoleak type III (General disorders) | 5 (6) | 5 (5) | 3 (3)
Unknown cause of death (General disorders) | 1 (1) | 4 (4) | 0 (0)
Vascular stent-graft occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Choledocholithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to antibiotic (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction to contrast agent (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Leg infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nosocomial pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Vascular graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Elbow fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fractured ethmoid (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intraoperative arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Advanced lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid rhinorrhoea (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Limb paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurological impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord ischemia (Nervous system disorders) | 0 (0) | 6 (6) | 0 (0)
Spinal subdural hematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Toxic metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device migration (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 2 (2) | 1 (1) | 0 (0)
Stent occlusion (Product Issues) | 1 (1) | 3 (3) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0)
Acute nonoliguric renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute on chronic renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Bladder paralysis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired renal function (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery dissection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal artery perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal function aggravated (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal hematoma (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Renal infarction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Retention urine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Dyspnea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute limb ischemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aneurysm enlargement (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic intramural hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortoiliac occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial bleeding (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Arterial rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Celiac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
External iliac artery perforation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral artery perforation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thoracic aneurysm, ruptured (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thoracic aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Type A aortic dissection (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Type B aortic dissection (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | fEVAR (N=92) | bEVAR (N=136) | fbEVAR (N=31)
Stent-graft endoleak type II (General disorders) | 6 (6) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT05143138/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT05143138/SAP_001.pdf